CLINICAL TRIAL: NCT05460169
Title: Effect of Renal Denervation in Hypertensive Patients With Autosomal Dominant Polycystic Kidney Disease
Brief Title: Renal Denervation in ADPKD- RDN-ADPKD Study
Acronym: RDN-ADPKD
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Erlangen-Nürnberg Medical School (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RDN2021ADPKD
Record Dates: First submitted 2022-06-15; First posted 2022-07-15 (Actual); Last update posted 2024-11-05 (Actual); Status verified 2024-11

CONDITIONS: Uncontrolled Hypertension; Autosomal Dominant Polycystic Kidney Disease; Renal Denervation
Keywords: Uncontrolled Hypertension; Autosomal Dominant Polycystic Kidney Disease; Renal denervation
MeSH Terms: conditions — Polycystic Kidney, Autosomal Dominant

STUDY DESIGN:
Intervention Model Description: RDN-ADPKD is a prospective, randomized (1:1, central randomization), single-centre, hypothesis-generating, feasibility study. Patients are randomized into I-RDN-group and D-RDN-group, respectively. After 3 months, patients in the D-RDN-group will undergo RDN-procedure and will be followed for additional 36 months. Hence, study design allows several comparisons both of whole study group (at same time-point of follow-up) as well as between I-RDN-group and D-RDN-group.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Immediate Renal Denervation Group (I-RDN-group) (Active Comparator): Patients are randomized into (immediate) I-RDN-group and (delayed) D-RDN-group, respectively. All subjects in the I-RDN-group will undergo a diagnostic, renal angiogram immediately (based on clinical grounds to rule out renal artery stenosis), which should be per Institutional practice via femoral artery access. Renal Denervation procedure will be applied using the Paradise® Renal Denervation System. The Paradise® Renal Denervation System is a catheter-based device designed to use ultrasound energy to thermally ablate the afferent and efferent nerves surrounding the renal artery and serving the kidney.
  Interventions: Device: Renal denervation
- Delayed Renal Denervation Group (D-RDN-group) (Other): 3 months after randomization, patients in the (delayed) D-RDN-group will undergo renal denervation procedure after undergoing a diagnostic, renal angiogram and will be followed for additional 36 months.
  Interventions: Device: Renal denervation

INTERVENTIONS:
Device: Renal denervation — The Paradise® Renal Denervation System (Paradise System) is CE-marked in countries accepting the CE mark. The system is a catheter-based device designed to use ultrasound energy to thermally ablate the afferent and efferent nerves surrounding the renal artery and serving the kidney.

SUMMARY:
RDN-ADPKD is a prospective, randomized (1:1, central randomization), single-center, hypothesis-generating, feasibility study. The purpose of the RDN-ADPKD study is to demonstrate efficacy and document safety of renal denervation (RDN) with the Paradise System in hypertensive patients with ADPKD.

DETAILED DESCRIPTION:
1. Introduction:Increased blood pressure (BP) is a common finding in patients with autosomal dominant polycystic kidney disease (ADPKD) which is one of the leading causes of end stage renal disease. Previously, it was shown that hypertensive patients with ADPKD have increased sympathetic nerve activity regardless of renal function. This was one of the pathogenetic mechanisms that leads to the progression of renal failure, even independent of BP. Recent clinical studies have indicated that invasive, catheter-based renal denervation (RDN) decreases sympathetic nerve activity. Up to date, only two single case reports have suggested a safe and effective procedure of RDN in an ADPKD patient with uncontrolled hypertension.
2. Study purpose: The purpose of the RDN-ADPKD pilot study is to demonstrate efficacy and document safety of RDN with the Paradise System in hypertensive patients with ADPKD.
3. Study design: RDN-ADPKD is a prospective, randomized (1:1, central randomization), single-center, hypothesis-generating, feasibility study.

   Patients are randomized into (immediate) I-RDN-group and (delayed) D-RDN-group, respectively. After 3 months, patients in the D-RDN-group will undergo RDN-procedure and will be followed for additional 36 months. Hence, study design allows several comparisons both of whole study group (at same time-point of follow-up) as well as between I-RDN-group and D-RDN-group.
4. Patient population: 44 hypertensive patients with ADPKD are randomized with 22 patients allocated to the I-RDN-group and 22 patients to the D-RDN-group (receiving RDN after 3 months), respectively.
5. Primary endpoint: The primary endpoint of this pilot study is the change in systolic 24-h ambulatory BP at 3 months post-procedure in the whole study group (irrespective whether treated immediate [I-RDN-group] or delayed [D-RDN-group]) compared to baseline.
6. Visit and Follow-Up Schedule: The primary objective will be assessed at 13 weeks (3 months) post-procedure in both groups. Scheduled in-clinic follow-up (FU) visits will occur at least at 13 (3 months) and 26 (6 months) 52 (12 months), 78 weeks (18 months),104 weeks (24 months), 130 weeks (30 months) and 156 weeks (36 months) post procedure; however, scheduled Follow-Up visits at 3, 7,20 weeks, 78 weeks and 130 weeks post-procedure are possible as in-clinic FU visit as well as ambulant visit at the allocation centre(s) of the referring physician.
7. Randomization: The subjects will be randomized to I-RDN group or D-RDN group at Visit 2.
8. Medication Adherence: Adherence to drug therapy will be captured by interviewing patients, checking the patient's BP diary and by urinary toxicological analysis at baseline, 26 weeks, 52 weeks, 104 weeks and 156 weeks post-procedure visit.
9. Safety Signals: A major combined safety endpoint is the incidence of any major adverse events (MAE) through the 36 months Follow-up.
10. Escape Criteria: Enrolled subjects will be excluded:

    * if home BP increases to ≥160 systolic or ≥100 mmHg diastolic pre-randomization, confirmed by office (attended) BP ≥170/105 mmHg will be excluded
    * if office (attended) BP exceeds ≥170/105 mmHg pre-randomization, confirmed by 7-day average of home BP measurements ≥ 160/100 mmHg (excluding white coat effect) or confirmed by office (attended) BP ≥170/105 mmHg at another study visit.
11. Ethics: The study will be conducted in accordance with the declaration of Helsinki, REGULATION (EU) 2017/745, EN ISO 14155:2020, FDA 21 CFR parts 50, 54, 56, 812 and other applicable local and national regulations.

ELIGIBILITY:
Inclusion Criteria:

* Patients with ADPKD
* Systolic office (attended) BP ≥130 mmHg or diastolic office (attended) BP ≥80 mmHg confirmed by 24-h ambulatory BP systolic ≥125 mmHg or diastolic ≥75 mmHg despite treatment with 1-4 drug classes (RAS blockade is mandatory, unless intolerance to RAS blockers has been documented) The rationale of these inclusion criteria reflect the November 2021 updated knowledge of RDN according to international consensus reports, in particular in face of conducting clinic studies and randomized controlled trials and does not necessarily reflect the current application of RDN in clinical practice). Moreover, the most recent updated KDIGO guidelines recommend a target office BP < 120 mmHg in patients with chronic kidney disease.1.
* Patient is adhering to a stable drug regimen without changes for a minimum of 4 weeks
* Individual is ≥ 18 years of age, both genders are included

Exclusion Criteria:

* eGFR < 40ml/min/1.73m² (according to the currently used estimation formulas: MDRD (Modification of Diet in Renal Disease), CKD-EPI (Chronic Kidney Disease Epidemiology Collaboration))
* Anatomically significant renal artery abnormality in either renal artery which in the eyes of the interventionalist would interfere with safe catheter placement
* Prior renal denervation procedure
* Office (attended) BP ≥180 mmHg systolic and/or ≥110 mmHg diastolic
* 24-h ambulatory BP ≥160 mmHg systolic
* Other cause of hypertension that can be treated by intervention/surgery (e.g. hemodynamically relevant renal artery stenosis, functional adrenal adenoma)
* Type 1 diabetes mellitus
* Proteinuria (>3g/g Kreatinin)
* Contraindication to MRI
* Individual has experienced a myocardial infarction, unstable angina pectoris, or a cerebrovascular accident within 3 months of the screening visit
* Subject is pregnant, nursing, or intends to become pregnant
* Enrollment in another interventional research protocol
* Any condition that, at the discretion of the investigator, would preclude participation in the study (e.g. non-adherence)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2022-06-14 (Actual); Primary Completion 2028-03 (Estimated); Study Completion 2028-03 (Estimated)

PRIMARY OUTCOMES:
change in systolic 24-h ambulatory BP [whole study group] | 3 months post-procedure
  change in systolic 24-h ambulatory BP at 3 months post-procedure from pre-treatment in the whole study group (irrespective whether treated immediate [I-RDN-group] or delayed [D-RDN-group]).

SECONDARY OUTCOMES:
Change in diastolic 24-h ambulatory BP [whole study group] | 3 months post-procedure
  Change in diastolic 24-h ambulatory BP at 3 months post-procedure in the whole study group (irrespetive whether treated immmediate (I-RDN-group) or delayed (D-RDN-group) compared to pre-treatment
Change in systolic and diastolic 24-h ambulatory BP [whole study group] | 6, 12, 18, 24, 30, 36 months post-procedure
  Change in systolic and diastolic 24-h ambulatory BP at 6, 12, 18, 24, 30 and 36 months post-procedure in the whole study group (irrespective whether treated immediate [I-RDN-group] or delayed [D-RDN-group]) compared to pre-treatment
Change in systolic and diastolic 24-h ambulatory BP [separate study groups] | 3 months post-procedure
  Change in systolic and diastolic 24-h ambulatory BP at 3 months post-procedure from pre-treatment in the I-RDN-group versus the change in systolic 24-h ambulatory BP prior procedure from pre-treatment in D-RDN-group
Responder rate in BP [separate study groups] | 3 months post-procedure
  Responder rate in BP (systolic office BP ≥ 5 mmHg, or 24-h systolic ambulatory BP ≥ 3 mmHg) at 3 months pre-treatment in the I-RDN-group versus responder rate in BP from pre-treatment to 3 months later in the D-RDN-group.
Change in systolic and diastolic office (attended) BP [whole study group] | 3, 6, 12, 18, 24, 30, 36 months post-procedure
  Change in systolic and diastolic office (attended) BP at 3, 6, 12, 18 and 24, 30, 36 months post-procedure in the whole study group compared to pre-treatment
Change in systolic and diastolic office (attended) BP [separate study groups] | 3 months post-procedure
  Change in systolic office (attended) BP at 3 months post-procedure from pre-treatment in the I-RDN-group versus the change prior procedure from pre-treatment in D-RDN-group
Change in systolic and diastolic home BP (IEM-Tel-O-Graph-GSM) [whole study group] | 3, 6, 12, 24 and 36 months post-procedure
  Change in systolic and diastolic home BP (IEM-Tel-O-Graph-GSM) at 3, 6, 12, 24 and 36 months post-procedure in the whole study group compared to pre-treatment
Change in systolic and diastolic home BP (IEM-Tel-O-Graph-GSM) [separate study groups] | 3 months post-procedure
  Change in systolic and diastolic home BP at 3 months post-procedure in the I-RDN-group versus the change prior procedure from pre-treatment in D-RDN-group.
Win ratio analysis (BP change and decrease of medication number) [separate study groups] | 3 months post-procedure
  Win ratio analysis will be conducted, with the criteria 24h ambulatory systolic BP change > 3 mmHg, office systolic BP change > 5 mmHg, and decrease of medication number from pre-treatment to 3 month post procedure in the I-RDN group versus pre-treatment to 3 months later in D-RDN-group.
Win ratio analysis (BP change and decrease of drug burden index ) [separate study groups] | 3 months post-procedure
  Win ratio analysis will be conducted, with the criteria 24h ambulatory systolic BP change > 3 mmHg, office systolic BP change > 5 mmHg, and any decrease of drug burden index from pre-treatment to 3 month post procedure in the I-RDN group versus pre-treatment to 3 months later in D-RDN-group.
Win ratio analysis (BP change and decrease of antihypertensive load index ) [separate study groups] | 3 months post-procedure
  Win ratio analysis will be conducted, with the criteria 24h ambulatory systolic BP change > 3 mmHg, office systolic BP change > 5 mmHg, and any decrease of antihypertensive load index from pre-treatment to 3 month post procedure in the I-RDN group versus pre-treatment to 3 months later in D-RDN-group
Change in serum creatinine derived estimated glomerular filtration rate (eGFR) [whole study group] | 3, 6, 12, 18 and 24, 30, 36 months post-procedure
  Change in serum creatinine derived estimated glomerular filtration rate (eGFR) at 3, 6, 12, 18 and 24, 30 and 36 months post-procedure in the whole study group compared to pre-treatment
Change in cystatin C derived eGFR [whole study group] | 3, 6, 12, 18 and 24, 30, 36 months post-procedure
  Change in cystatin C derived estimated glomerular filtration rate (eGFR) at 3, 6, 12, 18 and 24, 30, 36 months post-procedure in the whole study group compared to pre-treatment
Change in total kidney volume (assessed by magnetic resonance imaging) [whole study group] | 6, 12, 24, 36 months post-procedure
  Change in total kidney volume (assessed by magnetic resonance imaging) at 6, 12, 24, 36 months post-procedure in the whole study group compared to pre-treatment
Change in measured GFR (assessed by single-shot iohexol clearance) [whole study group] | 6, 12, 24, 36 months post-procedure
  Change in measured GFR (assessed by single-shot iohexol clearance) at 6, 12, 24 and 36 months post-procedure in the whole study group compared to pre-treatment
Change in proteinuria [whole study group] | 3, 6, 12, 18, 24, 30 and 36 months post-procedure
  Change in proteinuria (per g urinary creatinine) at 3, 6, 12, 18, 24, 30 and 36 months post-procedure from pre-treatment.
Change in albuminuria [whole study group] | 3, 6, 12, 18, 24, 30 and 36 months post-procedure
  Change in albuminuria (per g urinary creatinine) at 3, 6, 12, 18, 24, 30 and 36 months post-procedure from pre-treatment.
Change in urine sodium [whole study group] | 3, 6, 12, 18, 24, 30 and 36 months post-procedure
  Change in urine sodium (per g urinary creatinine) at 3, 6, 12, 18, 24, 30 and 36 months post-procedure from pre-treatment.
Change in urine potassium [whole study group] | 3, 6, 12, 18, 24, 30 and 36 months post-procedure
  Change in urine potassium (per urinary creatinine) at 3, 6, 12, 18, 24, 30 and 36 months post-procedure from pre-treatment.
Change in urine creatinine concentration [whole study group] | 3, 6, 12, 18, 24, 30 and 36 months post-procedure
  Change in urine creatinine concentration at 3, 6, 12, 18, 24, 30 and 36 months post-procedure from pre-treatment.
Change of the slope of eGFR [whole study group] | 3, 6, 12, 18, 24, 30 and 36 months post-procedure
  Change of the slope of eGFR after 3, 6, 12, 18, 24, 30 and 36 months post-procedure from pre-treatment compared to the historical slope the year before in the total study group.
Change in serum creatinine derived eGFR [separate study groups] | 3 months post-procedure
  Change in serum creatinine derived eGFR at 3 months post-procedure from pre-treatment in the I-RDN-group versus the change prior procedure from pre-treatment in D-RDN-group
Change in cystatin C derived eGFR [separate study groups] | 3 months post-procedure
  Change in cystatin C derived eGFR at 3, 6, 12, 18 and 24, 30, 36 months post-procedure from pre-treatment in the I-RDN-group versus the change prior procedure from pre-treatment in D-RDN-group
Change in proteinuria [separate study groups] | 3 months post-procedure
  Change in proteinuria from pre-procedure pre-treatment in the I-RDN-group versus the change from pre-treatment to 3 months later in the D-RDN-group.
Change in albuminuria [separate study groups] | 3 months post-procedure
  Change in albuminuria from pre-procedure pre-treatment in the I-RDN-group versus the change from pre-treatment to 3 months later in the D-RDN-group.
Change in urine sodium [separate study groups] | 3 months post-procedure
  Change in urine sodium from pre-procedure pre-treatment in the I-RDN-group versus the change from pre-treatment to 3 months later in the D-RDN-group.
Change in urine potassium [separate study groups] | 3 months post-procedure
  Change in urine potassium from pre-procedure pre-treatment in the I-RDN-group versus the change from pre-treatment to 3 months later in the D-RDN-group.
Change in urine creatinine concentration [separate study groups] | 3 months post-procedure
  Change in urine creatinine concentration from pre-procedure pre-treatment in the I-RDN-group versus the change from pre-treatment to 3 months later in the D-RDN-group.
Change of the slope of eGFR [separate study groups] | 3 month post-procedure
  Change of the slope of eGFR after 3 month post-procedure from pre-treatment (including eGFR values) in the I-RDN group compared to change after 3 month FU from pre-treatment in the D-RDN group.
Level of pain (related to autosomal dominant polycystic kidney disease) determined by the use of a visual analogue scale [whole study group] | 3, 6, 12, 24, 36 months post-procedure
  Level of pain (related to autosomal dominant polycystic kidney disease) determined by the use of a visual analogue scale (minimum value=0, representing no pain; maximum value=100, representing most imaginable pain) at 3, 6, 12, 24, 36 months post-procedure in the whole study group compared to pre-treatment.
Change in Quality of life (QoL) (e.g. EQ-5D-5L) [whole study group] | 3, 6, 12, 24 and 36 months post-procedure
  Change in Quality of life (QoL) (e.g. EQ-5D-5L; minimum value=0, representing best imaginable health status; maximum value=100, representing worst imaginable health status) at 3, 6, 12, 24 and 36 months post-procedure in the whole study group compared to pre-treatment
Change in plasma and urinary biomarkers (e.g. albumin, copeptin) | 6, 12 months post-procedure
  Change in plasma and urinary biomarkers (e.g. albumin, copeptin) at 6, 12 months post-procedure in the whole study group compared to pre-treatment

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital FAU Erlangen-Nürnberg, Erlangen, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] St Pierre K, Cashmore BA, Bolignano D, Zoccali C, Ruospo M, Craig JC, Strippoli GF, Mallett AJ, Green SC, Tunnicliffe DJ. Interventions for preventing the progression of autosomal dominant polycystic kidney disease. Cochrane Database Syst Rev. 2024 Oct 2;10(10):CD010294. doi: 10.1002/14651858.CD010294.pub3. PMID 39356039

DOCUMENTS (1):
  • Statistical Analysis Plan (2023-11-17): https://cdn.clinicaltrials.gov/large-docs/69/NCT05460169/SAP_000.pdf